CLINICAL TRIAL: NCT00192504
Title: A Phase 1, Randomized, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of a Single Intravenous Dose of MEDI-524, a Humanized Enhanced Potency Monoclonal Antibody to Respiratory Syncytial Virus (RSV), in Otherwise Healthy Children Hospitalized With RSV Infection
Brief Title: Safety Study of a Monoclonal Antibody to Respiratory Syncytial Virus (RSV) in Children Hospitalized With RSV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Genevieve A. Losonsky, MD/Vice President, Clinical Development, MedImmune, LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MI-CP106
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Results first posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2006-10

CONDITIONS: Respiratory Syncytial Virus Prophylaxis
Keywords: MEDI-524; Motavizumab; respiratory syncytial virus; children; intravenous; Rezield
MeSH Terms: interventions — motavizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Motavizumab, 3 mg/kg as a single intravenous dose (Experimental): Motavizumab, 3 mg/kg as a single intravenous dose administered on Day 0
  Interventions: Biological: Motavizumab
- Motavizumab, 15 mg/kg as a single intravenous dose (Experimental): Motavizumab, 15 mg/kg as a single intravenous dose administered on Day 0
  Interventions: Biological: Motavizumab
- Motavizumab, 30 mg/kg as a single intravenous dose (Experimental): Motavizumab, 30 mg/kg as a single intravenous dose administered on Day 0
  Interventions: Biological: Motavizumab
- Placebo, as a single intravenous dose (Placebo Comparator): Placebo, as a single intravenous dose administered on Day 0
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Motavizumab — Single dose of Motavizumab at a dose of 3 mg/kg administered intravenously (in the vein) on Day 0
  Other Names: MEDI-524
  Arms: Motavizumab, 3 mg/kg as a single intravenous dose
Biological: Motavizumab — Single dose of Motavizumab at a dose of 15 mg/kg administered intravenously (in the vein) on Day 0
  Other Names: MEDI-524
  Arms: Motavizumab, 15 mg/kg as a single intravenous dose
Biological: Motavizumab — Single dose of Motavizumab at a dose of 30 mg/kg administered intravenously (in the vein) on Day 0
  Other Names: MEDI-524
  Arms: Motavizumab, 30 mg/kg as a single intravenous dose
Other: Placebo — Single dose of placebo administered intravenously (in the vein) on Day 0
  Arms: Placebo, as a single intravenous dose

SUMMARY:
The purpose of this study is to determine the safety of motavizumab (MEDI-524) following a single intravenous dose in children hospitalized with respiratory syncytial virus (RSV).

DETAILED DESCRIPTION:
This study was designed as a Phase 1, randomized, double-blind, placebo-controlled, dose-escalation, multicenter clinical study to evaluate the safety, tolerability, serum concentrations, and immunogenicity of a single intravenous dose of motavizumab (MEDI-524) and the effect on the amount of respirtory syncytial virus (RSV) in the respiratory tract (nasopharynx) of otherwise healthy children hospitalized with RSV infection.

ELIGIBILITY:
Inclusion Criteria:

* Previously healthy
* Age 24 months and younger at the time of randomization
* Gestational age of 36 weeks gestation and older
* Randomization within 24 hours after hospitalization
* Hospitalized for lower respiratory tract illness (ie, respiratory syncytial virus (RSV) bronchiolitis and/or pneumonia) documented by positive RSV antigen detection or culture in respiratory secretions within 72 hours before randomization

Exclusion Criteria:

* Already received or would receive ribavirin or other anti-viral treatment for the current episode of RSV infection prior to randomization
* Required intubation for ventilatory support
* Any medically significant underlying ongoing chronic illness or organ system dysfunction or other known acute illness, other than RSV infection
* Known renal impairment, hepatic dysfunction, hematologic abnormalities, seizure or other neurologic disorder or immunodeficiency
* Requirement for supplemental oxygen at any time prior to the current RSV infection (brief use of oxygen in the immediate postnatal period to treat a transient condition was allowed)
* Mechanical ventilation at any time prior to the onset of the current RSV infection
* Congenital heart disease (children with medically or surgically corrected patent ductus arteriosus [PDA], small atrial septal defect [ASD] or ventricular septal defect [VSD] were allowed)
* Previous reaction to intravneous immunoglobulin (IVIG), blood products, or other foreign proteins
* Prior use of IVIG, RSV-IGIV (RespiGam), palivizumab (Synagis), or other immunoglobulin products within the past 2 months
* Currently receiving other investigational agents or have received any other investigational agents within the last 3 months
* Prior or current participation in any investigational study with a therapeutic agent or vaccine for RSV

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2004-03; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve A Losonsky, MD, Study Director — MedImmune LLC

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The screening period occurred within 24 hours before randomization. All subjects who were screened were randomized into the study.
Groups:
- Motavizumab (MEDI-524), 3 mg/kg: Motavizumab, 3 mg/kg as a single intravenous dose administered on Day 0
- Motavizumab (MEDI-524), 15 mg/kg: Motavizumab, 15 mg/kg as a single intravenous dose administered on Day 0
- Motavizumab (MEDI-524), 30 mg/kg: Motavizumab, 30 mg/kg as a single intravenous dose administered on Day 0
- Placebo: Placebo, as a single intravenous dose administered on Day 0
Period: Overall Study
Arm/Group | Motavizumab (MEDI-524), 3 mg/kg | Motavizumab (MEDI-524), 15 mg/kg | Motavizumab (MEDI-524), 30 mg/kg | Placebo
Started | 5 | 5 | 6 (Baseline demographics are not available on one patient who did not receive study drug.) | 15
Completed | 4 | 5 | 5 | 15
Not Completed | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Dosing window missed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motavizumab (MEDI-524), 3 mg/kg | Motavizumab (MEDI-524), 15 mg/kg | Motavizumab (MEDI-524), 30 mg/kg | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: months] — Age at randomization
  months | 8.84 (6.62) | 3.18 (1.56) | 10.78 (9.07) | 7.43 (7.69) | 7.51 (7.19)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline demographics are not available for one patient in the 30 mg/kg group because the patient received no study drug in the study.
  Participants
    Female | 2 | 4 | 1 | 3 | 10
    Male | 3 | 1 | 4 | 12 | 20
Race/Ethnicity, Customized [Number; unit: Participants]
  White/Non-Hispanic | 1 | 0 | 1 | 1 | 3
  Hispanic | 4 | 5 | 4 | 14 | 27
Region of Enrollment [Number; unit: participants]
  Chile | 4 | 5 | 4 | 14 | 27
  United States | 1 | 0 | 1 | 1 | 3
Weight [Mean (Standard Deviation); unit: Kilograms] | 8.728 (1.392) | 5.516 (0.891) | 9.194 (3.43) | 7.386 (3.218) | 7.599 (2.903)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Adverse Events Through 30 Days After Dosing
Description: Safety and tolerability of motavizumab (MEDI-524) was measured by adverse events through 30 days after dosing
Time Frame: From the start of treatment to 30 days after dosing
Population: All patients who recieved study drug were included in the analysis of safety.
Measure: Number; unit: Participants
Arm/Group | Motavizumab (MEDI-524), 3 mg/kg | Motavizumab (MEDI-524), 15 mg/kg | Motavizumab (MEDI-524), 30 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 15
Participants | 3 | 5 | 3 | 6

2. Primary Outcome: Number of Subjects Reporting Serious Adverse Events Through 30 Days After Dosing
Description: Safety and tolerability of motavizumab (MEDI-524) was measured by serious adverse events through 30 days after dosing
Time Frame: From the start of treatment to 30 days after dosing
Measure: Number; unit: participants
Arm/Group | Motavizumab (MEDI-524), 3 mg/kg | Motavizumab (MEDI-524), 15 mg/kg | Motavizumab (MEDI-524), 30 mg/kg | Placebo
Number analyzed (Participants) | 4 | 5 | 5 | 15
participants | 0 | 0 | 1 | 1

3. Secondary Outcome: To Describe the Immunogenicity of Motavizumab (MEDI-524) Following a Single IV Dose at Day 0
Description: The serum anti-motavizumab antibody titers were measured in subjects on Day 0 (before dosing). Anti-motavizumab antibody assays were performed at MedImmune using a qualified assay.
Time Frame: Immediately before dosing on Day 0
Population: All patients who received a full dose of study drug were included in the analysis of immunogenicity.
Measure: Number; unit: Participants
Arm/Group | Motavizumab (MEDI-524), 3 mg/kg | Motavizumab (MEDI-524), 15 mg/kg | Motavizumab (MEDI-524), 30 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 15
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: To Describe the Immunogenicity of Motavizumab (MEDI-524) Following a Single IV Dose at Day 30
Description: The serum anti-motavizumab antibody titers were measured in subjects on Day 30. Anti-motavizumab antibody assays were performed at MedImmune using a qualified assay.
Time Frame: Day 30
Population: All patients who received a full dose of study drug were included in the analysis of immunogenicity. One patient in the 3 mg/kg group was not assessed for immunogenicity.
Measure: Number; unit: Participants
Arm/Group | Motavizumab (MEDI-524), 3 mg/kg | Motavizumab (MEDI-524), 15 mg/kg | Motavizumab (MEDI-524), 30 mg/kg | Placebo
Number analyzed (Participants) | 4 | 5 | 5 | 15
Participants | 0 | 0 | 0 | 0

5. Primary Outcome: The Occurrence of Increased Toxixity Grade From Baseline as Determined by Laboratory Evaluations
Description: Safety and tolerability of motavizumab (MEDI-524) was measured by the occurrence of increased toxicity grade from baseline as determined by laboratory evaluations (complete blood count, aspartate aminotransferase (AST), alanine aminotransferase (ALT), blood urea nitrogen (BUN), creatinine, and urinalysis) at baseline and at each study collection time point following dosing
Time Frame: From the start of treatment to 30 days after dosing
Population: All patients who recieved study drug were included in the analysis of safety.
Measure: Number; unit: Participants
Arm/Group | Motavizumab (MEDI-524), 3 mg/kg | Motavizumab (MEDI-524), 15 mg/kg | Motavizumab (MEDI-524), 30 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 15
Participants | 0 | 1 | 1 | 1

6. Primary Outcome: To Describe the Mean Trough Serum Concentrations of Motavizumab (MEDI-524) Administered as a Single Intravenous Dose at Day 2 and Day 30
Description: Mean trough serum concentrations of motavizumab (MEDI-524) were collected on Day 2 and on Day 30. Serum concentrations of MEDI-524 were analysed using a qualified enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 2 and Day 30
Population: All patients who recieved a full dose of study drug were included in the analysis of trough serum concentrations. One patient in the 3 mg/kg group was not assessed for serum trough levels at either Day 2 or Day 30.
Measure: Mean (Standard Deviation); unit: Micrograms per mililiter
Arm/Group | Motavizumab (MEDI-524), 3 mg/kg | Motavizumab (MEDI-524), 15 mg/kg | Motavizumab (MEDI-524), 30 mg/kg | Placebo
Number analyzed (Participants) | 4 | 5 | 5 | 15
Micrograms per mililiter
  Trough Serum Concentration at Day 2 | 61.78 (20.09) | 170.8 (38.43) | 333.2 (99.86) | 0 (0)
  Trough Serum Concentration at Day 30 | 16.63 (13.08) | 59.18 (12.72) | 80.28 (27.34) | 0 (0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of the first administration of motavizumab (MEDI-524) to 30 days after dosing.
Arm/Group | Motavizumab (MEDI-524), 3 mg/kg | Motavizumab (MEDI-524), 15 mg/kg | Motavizumab (MEDI-524), 30 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 1/5 | 1/15
Other Adverse Events (participants affected / at risk) | 3/5 | 5/5 | 3/5 | 6/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motavizumab (MEDI-524), 3 mg/kg (N=5) | Motavizumab (MEDI-524), 15 mg/kg (N=5) | Motavizumab (MEDI-524), 30 mg/kg (N=5) | Placebo (N=15)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motavizumab (MEDI-524), 3 mg/kg (N=5) | Motavizumab (MEDI-524), 15 mg/kg (N=5) | Motavizumab (MEDI-524), 30 mg/kg (N=5) | Placebo (N=15)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Disbacteriosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemodynamic instability (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemophilus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Heat rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superinfection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.